CLINICAL TRIAL: NCT06240585
Title: Gastroparesis as an Early Sign of Sepsis
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0027-24-MMC
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Gastroparesis and Sepsis
MeSH Terms: conditions — Gastroparesis; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with ICU-acquired bacteremia
  Interventions: Other: presence of gastroparesis as an early sign for sepsis (bacteremia)- measurement of gastric residual volume
- patients without ICU-acquired bacteremia

INTERVENTIONS:
Other: presence of gastroparesis as an early sign for sepsis (bacteremia)- measurement of gastric residual volume — presence of gastroparesis as an early sign for sepsis (bacteremia)-measurement of gastric residual volume
  Groups: patients with ICU-acquired bacteremia

SUMMARY:
Upper gastrointestinal tract disorders, such as gastroparesis, are common in critically ill patients in the ICU, estimated at 60%. Gastroparesis symptoms include nausea, vomiting and abdominal pain. Risk factors for the development of gastroparesis include diabetes, surgical injury to the vagus nerve (such as certain types of bariatric surgery, and in the past - surgeries for patients who suffered from peptic ulcer), use of drugs that inhibit the activity of the digestive system such as opiates, anticholinergic drugs, sepsis, as well as being bedridden and inactive - are all common conditions in critically ill patients.

There are different definitions for gastroparesis. One of the accepted definitions refers to gastric residual volume (GRV) over 200 ml at one measurement. Gastroparesis is found in some studies to be associated with increased morbidity and mortality in critically ill patients. As mentioned above, it is known that sepsis is a risk factor for gastroparesis. According to our experience based on treatment of a large number of septic patients, we have the impression that often gastroparesis is an early sign for the development of sepsis. We did not find any studies that tested this hypothesis.

In this study we would like to investigate whether the development of gastroparesis in critical patients in intensive care can be a predictive sign for the development of sepsis.

ELIGIBILITY:
Inclusion Criteria: Patients aged 18--99 who were admitted to the general intensive care unit from January 2015 to April 2021, and who were diagnosed with acquired bacteremia in the ICU (positive blood culture after 48 hours or more from ICU admission). As a control group we will collect data regarding a similar number of patients who were admitted during this time period but were not diagnosed with acquired bacteremia or sepsis during their stay in the unit.

-

Exclusion Criteria: Patients who did not meet the above criteria or for whom data were missing. Likewise, patients who did not have a nasogastric tube will be excluded (we cannot test gastirc residual volume) as well as patients who were admitted after abdominal surgery (gastroparesis is a common finding in these patients regardless of sepsis and may be a confounder. In addition, acquired bacteremia in these patients could be the result of a surgical complication, such as intra-abdominal sepsis secondary to intestinal leak etc., and gastroparesis usually accompanies abdominal sepsis and will not be the result of sepsis per-se).

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acquired ICU bacteremia
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
gastroparesis as an early sign for sepsis (bacteremia) | 24 hours before appearance of bacteremia

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided